CLINICAL TRIAL: NCT01768741
Title: A Randomized Controlled Trial of Laparoscopic Versus Open Liver Resection in the Treatment of Hepatocellular Carcinoma
Brief Title: Laparoscopic Versus Open Liver Resection in the Treatment of Hepatocellular Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Xiujun Cai, Executive Vice-President, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SRRSH20121225-2
Record Dates: First submitted 2013-01-13; First posted 2013-01-15 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Laparoscopic liver resection group (Active Comparator)
  Interventions: Procedure: Laparoscopic liver resection
- Open liver resection (Active Comparator)
  Interventions: Procedure: Open liver resection

INTERVENTIONS:
Procedure: Laparoscopic liver resection — participants will be performed with laparoscopic hepatectomy using laparoscopic instruments
  Other Names: Laparoscopic hepatectomy
  Arms: Laparoscopic liver resection group
Procedure: Open liver resection — participants will be performed with open hepatectomy using laparotomic instruments
  Other Names: Open hepatectomy
  Arms: Open liver resection

SUMMARY:
The purpose of this study is to investigate the clinical value of laparoscopic liver resection in the treatment of hepatocellular carcinoma by assessing its Surgical and oncologic outcomes comparing with open liver resection.

ELIGIBILITY:
Inclusion Criteria:

* Liver solid tumor, with clinical diagnosis of hepatocellular carcinoma
* Located at segment Ⅱ、Ⅲ、Ⅳb、Ⅴ or Ⅵ
* The tumor location and size do not affect the dissection of hepatic hilar region
* Tumor size less than 10cm
* Without portal vein tumor thrombus
* Without intrahepatic or distant metastasis
* Willingness to participate in the study
* Able to understand the nature of the study and what will be required of them
* Body mass index of between 18 and 35
* Child-Pugh classification of A to B
* American Society of Anesthesiologists (ASA) grading of I to III

Exclusion Criteria:

* Pregnant or lactating women
* Unwillingness to participate
* Inability to give written informed consent
* Child-Pugh classification of C
* ASA grading of IV to V
* Tumor invasion of the inferior vena cava or confluence part of hepatic vein
* Decompensated liver cirrhosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2012-12; Primary Completion 2016-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Total survival time and disease free survival time | up to 5 years

SECONDARY OUTCOMES:
Surgical margins | 7 days
Time to functional recovery | participants will be followed for the duration of hospital stay, an expected average of 6 days
Postoperative hospital stay | participants will be followed for the duration of hospital stay, an expected average of 7 days
Morbidity and mortality | up to 3 months
Quality of life | up to 1 year
Intraoperative parameters including operation time,pneumoperitoneum time, liver resection time, estimated blood loss,transfusion, as well as number,size and location of the tumor | participants will be followed for the duration of operation, an expected average of 90 min
Regulatory T cells and associated cytokines in peripheral blood | up to 5 years
  Regulatory T cells and associated cytokines in peripheral blood will be tested 1day before operation,5 days, 3,6 months and 1,3,5 years after operation
Regulatory T cells and associated cytokines in liver cancer、para-carcinoma and healthy liver tissue | 7 days

OTHER OUTCOMES:
Hospital costs | participants will be followed for the duration of hospital stay, an expected average of 9 days

CONTACTS AND LOCATIONS:
Overall Officials: Xiujun Cai, MD, Principal Investigator — Sir Run Run Shaw Hospital
Locations (1):
- Department of General Surgery, Institute of Minimally Invasive Surgery, Sir Run Run Shaw Hospital, Hangzhou, Zhejiang, China